CLINICAL TRIAL: NCT00000560
Title: Beta-Blocker Evaluation in Survival Trial (BEST)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double
Other Study IDs: 104
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2005-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Heart Failure, Congestive; Heart Failure
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Heart Failure | interventions — Adrenergic beta-Antagonists

INTERVENTIONS:
Drug: adrenergic beta antagonists

SUMMARY:
To determine if addition of a beta-blocker to standard therapy in Class III and Class IV heart failure patients reduced total mortality.

DETAILED DESCRIPTION:
BACKGROUND:

Controlled and uncontrolled studies suggested that beta-blockade improves ventricular function in congestive heart failure. Several trials suggested that beta-blockers may also reduce mortality. In the Beta-Blocker Heart Attack Trial, patients with a history of heart failure had less cardiac and sudden-death mortality than those who did not. Patients with a low ejection fraction in the Cardiac Arrhythmia Suppression Trial who were treated with beta-blockade also had a reduction in mortality. The Metoprolol in Dilated Cardiomyopathy trial randomized patients with dilated cardiomyopathies to treatment with metoprolol or placebo. There was a trend toward reduction in a morbidity and mortality endpoint in patients treated with metoprolol, but this was due entirely to a reduction in the need for cardiac transplantation. Thus, despite a reasonable theoretical basis and suggestive clinical studies, the concept that beta-blockers reduced mortality in congestive heart failure patients was unproved.

DESIGN NARRATIVE:

Randomized, double-blind, multicenter. Patients were assigned to standard therapy plus the addition of a beta-blocker (bucindolol) versus a placebo. The primary endpoint was total mortality. A radionuclide ventriculogram was performed within 60 days of randomization. History, physical examination, clinical laboratory studies, chest x-ray, electrocardiogram, and plasma norepinephrine levels were obtained within 14 days of randomization. Patients were stratified by hospital, congestive heart failure etiology, ejection fraction, and gender, and were assigned to a treatment group by an adaptive balancing scheme ("biased coin" randomization). Patients were randomized to either placebo plus standard congestive heart failure treatment or to the beta-blocker plus standard congestive heart failure treatment and followed for a minimum of 18 months. The over three year recruitment period began in May 1995 at the first 35 sites. An additional 55 sites began recruitment on August 14, 1995. Recruitment ended in December, 1998 with the enrollment of 2,708 patients.

ELIGIBILITY:
Men and women, ages 18 and over. Patients had compensated congestive heart failure due to idiopathic dilated cardiomyopathy or coronary disease with ejection fraction less than or equal to 0.35, were in the New York Heart Association functional class III or IV, and were taking an angiotensin-converting enzyme inhibitor, digitalis, and if needed, a diuretic. Patients with a specific indication for, or contraindication to, beta-blockade were excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1994-06; Study Completion 1999-09

CONTACTS AND LOCATIONS:
Overall Officials: Philip Lavori — Veterans Administration Hospital

REFERENCES:
- [Background] Design of the Beta-Blocker Evaluation Survival Trial (BEST). The BEST Steering Committee. Am J Cardiol. 1995 Jun 15;75(17):1220-3. doi: 10.1016/s0002-9149(99)80766-8. PMID 7778543
- [Background] Beta-Blocker Evaluation of Survival Trial Investigators; Eichhorn EJ, Domanski MJ, Krause-Steinrauf H, Bristow MR, Lavori PW. A trial of the beta-blocker bucindolol in patients with advanced chronic heart failure. N Engl J Med. 2001 May 31;344(22):1659-67. doi: 10.1056/NEJM200105313442202. PMID 11386264
- [Background] Aranda JM, Krause-Steinrauf HJ, Greenberg BH, Heng MK, Kosolcharoen PK, Renlund DG, Thaneemit-Chen S, White M, Cintron GB. Comparison of the beta blocker bucindolol in younger versus older patients with heart failure. Am J Cardiol. 2002 Jun 1;89(11):1322-6. doi: 10.1016/s0002-9149(02)02339-1. No abstract available. PMID 12031741
- [Background] Anderson JL, Krause-Steinrauf H, Goldman S, Clemson BS, Domanski MJ, Hager WD, Murray DR, Mann DL, Massie BM, McNamara DM, Oren R, Rogers WJ; Beta-Blocker Evaluation of Survival Trial (BEST) Investigators. Failure of benefit and early hazard of bucindolol for Class IV heart failure. J Card Fail. 2003 Aug;9(4):266-77. doi: 10.1054/jcaf.2003.42. PMID 13680547
- [Background] Domanski M, Krause-Steinrauf H, Deedwania P, Follmann D, Ghali JK, Gilbert E, Haffner S, Katz R, Lindenfeld J, Lowes BD, Martin W, McGrew F, Bristow MR; BEST Investigators. The effect of diabetes on outcomes of patients with advanced heart failure in the BEST trial. J Am Coll Cardiol. 2003 Sep 3;42(5):914-22. doi: 10.1016/s0735-1097(03)00856-8. PMID 12957443
- [Background] Eichhorn EJ, Grayburn PA, Mayer SA, St John Sutton M, Appleton C, Plehn J, Oh J, Greenberg B, DeMaria A, Frantz R, Krause-Steinrauf H. Myocardial contractile reserve by dobutamine stress echocardiography predicts improvement in ejection fraction with beta-blockade in patients with heart failure: the Beta-Blocker Evaluation of Survival Trial (BEST). Circulation. 2003 Nov 11;108(19):2336-41. doi: 10.1161/01.CIR.0000097111.00170.7B. Epub 2003 Nov 3. PMID 14597587
- [Background] Ghali JK, Krause-Steinrauf HJ, Adams KF, Khan SS, Rosenberg YD, Yancy CW, Young JB, Goldman S, Peberdy MA, Lindenfeld J. Gender differences in advanced heart failure: insights from the BEST study. J Am Coll Cardiol. 2003 Dec 17;42(12):2128-34. doi: 10.1016/j.jacc.2003.05.012. PMID 14680739
- [Background] Lindenfeld J, Ghali JK, Krause-Steinrauf HJ, Khan S, Adams K, Goldman S, Peberdy MA, Yancy C, Thaneemit-Chen S, Larsen RL, Young J, Lowes B, Rosenberg YD; BEST Investigators. Hormone replacement therapy is associated with improved survival in women with advanced heart failure. J Am Coll Cardiol. 2003 Oct 1;42(7):1238-45. doi: 10.1016/s0735-1097(03)00938-0. PMID 14522488
- [Background] Bristow MR, Krause-Steinrauf H, Nuzzo R, Liang CS, Lindenfeld J, Lowes BD, Hattler B, Abraham WT, Olson L, Krueger S, Thaneemit-Chen S, Hare JM, Loeb HS, Domanski MJ, Eichhorn EJ, Zelis R, Lavori P. Effect of baseline or changes in adrenergic activity on clinical outcomes in the beta-blocker evaluation of survival trial. Circulation. 2004 Sep 14;110(11):1437-42. doi: 10.1161/01.CIR.0000141297.50027.A4. Epub 2004 Aug 30. PMID 15337700
- [Background] O'Connor CM, Gottlieb S, Bourque JM, Krause-Steinrauf H, Anand I, Anderson JL, Plehn JF, Silver MA, White M, Carson P; BEST Investigators. Impact of nonfatal myocardial infarction on outcomes in patients with advanced heart failure and the effect of bucindolol therapy. Am J Cardiol. 2005 Mar 1;95(5):558-64. doi: 10.1016/j.amjcard.2004.11.001. PMID 15721091
- [Background] Grayburn PA, Appleton CP, DeMaria AN, Greenberg B, Lowes B, Oh J, Plehn JF, Rahko P, St John Sutton M, Eichhorn EJ; BEST Trial Echocardiographic Substudy Investigators. Echocardiographic predictors of morbidity and mortality in patients with advanced heart failure: the Beta-blocker Evaluation of Survival Trial (BEST). J Am Coll Cardiol. 2005 Apr 5;45(7):1064-71. doi: 10.1016/j.jacc.2004.12.069. PMID 15808765
- [Derived] Kristensen SL, Rorth R, Jhund PS, Shen L, Lee MMY, Petrie MC, Kober L, McMurray JJV; BEST Investigators. Microvascular complications in diabetes patients with heart failure and reduced ejection fraction-insights from the Beta-blocker Evaluation of Survival Trial. Eur J Heart Fail. 2018 Nov;20(11):1549-1556. doi: 10.1002/ejhf.1201. Epub 2018 May 4. PMID 29727039
- [Derived] Shen L, Jhund PS, Mogensen UM, Kober L, Claggett B, Rogers JK, McMurray JJV. Re-Examination of the BEST Trial Using Composite Outcomes, Including Emergency Department Visits. JACC Heart Fail. 2017 Aug;5(8):591-599. doi: 10.1016/j.jchf.2017.04.005. PMID 28774394
- [Derived] Breathett K, Allen LA, Udelson J, Davis G, Bristow M. Changes in Left Ventricular Ejection Fraction Predict Survival and Hospitalization in Heart Failure With Reduced Ejection Fraction. Circ Heart Fail. 2016 Oct;9(10):e002962. doi: 10.1161/CIRCHEARTFAILURE.115.002962. PMID 27656000
- [Derived] Jones LG, Sin MK, Hage FG, Kheirbek RE, Morgan CJ, Zile MR, Wu WC, Deedwania P, Fonarow GC, Aronow WS, Prabhu SD, Fletcher RD, Ahmed A, Allman RM. Characteristics and outcomes of patients with advanced chronic systolic heart failure receiving care at the Veterans Affairs versus other hospitals: insights from the Beta-blocker Evaluation of Survival Trial (BEST). Circ Heart Fail. 2015 Jan;8(1):17-24. doi: 10.1161/CIRCHEARTFAILURE.114.001300. Epub 2014 Dec 5. PMID 25480782
- [Derived] Aleong RG, Sauer WH, Davis G, Bristow MR. New-onset atrial fibrillation predicts heart failure progression. Am J Med. 2014 Oct;127(10):963-71. doi: 10.1016/j.amjmed.2014.06.006. Epub 2014 Jun 12. PMID 24931393
- [Derived] Aleong RG, Sauer WH, Davis G, Murphy GA, Port JD, Anand IS, Fiuzat M, O'Connor CM, Abraham WT, Liggett SB, Bristow MR. Prevention of atrial fibrillation by bucindolol is dependent on the beta(1)389 Arg/Gly adrenergic receptor polymorphism. JACC Heart Fail. 2013 Aug;1(4):338-344. doi: 10.1016/j.jchf.2013.04.002. PMID 24159564
- [Derived] O'Connor CM, Fiuzat M, Carson PE, Anand IS, Plehn JF, Gottlieb SS, Silver MA, Lindenfeld J, Miller AB, White M, Walsh R, Nelson P, Medway A, Davis G, Robertson AD, Port JD, Carr J, Murphy GA, Lazzeroni LC, Abraham WT, Liggett SB, Bristow MR. Combinatorial pharmacogenetic interactions of bucindolol and beta1, alpha2C adrenergic receptor polymorphisms. PLoS One. 2012;7(10):e44324. doi: 10.1371/journal.pone.0044324. Epub 2012 Oct 10. PMID 23071495
- Available data/document: Individual Participant Data Set: BEST — http://biolincc.nhlbi.nih.gov/studies/best/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol — http://biolincc.nhlbi.nih.gov/studies/best/
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/best/